CLINICAL TRIAL: NCT07056374
Title: Adaptive Anastomosis for Anterior Resection in Sigmoid and Proximal Rectal Cancer or Premalignant Lesion: a Multicentre Non-randomised Clinical Effectiveness Trial )ADAPT
Brief Title: Adaptive Anastomosis for Anterior Resection in Sigmoid and Proximal Rectal Cancer or Premalignant Lesions
Acronym: ADAPT
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Carponovum AB (Industry)
Responsible Party: Principal Investigator, Roel Hompes, MD, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: NL88846.018.25
Record Dates: First submitted 2025-04-17; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer; Sigmoid Cancer; Premalignant Lesion; Colorectal Cancer
Keywords: Anterior Resection; Adaptive anastomosis; Compression anastomosis; Anastomotic Leakage; Sigmoid resection; Partial Mesorectal Excision
MeSH Terms: conditions — Rectal Neoplasms; Sigmoid Neoplasms; Colorectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intervention C-REX RectoAid Cath: Patients with cancer of the sigmoid colon or proximal rectum, or premalignant lesions not amenable to endoscopic resection, that require elective anterior resection as the procedure of choice. The anastomosis will be created using an adaptive anastomosis technique using the C-REX RectoAid Cath.
  Interventions: Device: C-REX RectoAid Cath

INTERVENTIONS:
Device: C-REX RectoAid Cath — Adaptive anastomotis

SUMMARY:
Background: Anastomotic leakage (AL) after colorectal surgery remains a significant challenge, associated with increased morbidity, mortality, poor oncological outcomes, and reduced quality of life. Despite surgical advances, AL rates for colorectal procedures continue to range from 3% to 25%, especially in distal anastomoses.

The commonly used cross-stapled circular anastomosis for anterior resections (AR) activates a foreign body response delaying gastrointestinal wound healing and potentially increasing the risk of AL. Additionally, crossed stapler lines further increase the risk of AL. An adaptive anastomosis technique eliminates permanent foreign body material, thereby reducing negative effects on wound healing and avoiding cross-stapling potentially lowering the incidence of AL. These areas have shown to have a lower burst pressure compared to a single stapled anastomosis.

An adaptive anastomotic technique eliminates cross-stapling and permanent foreign body material in the anastomosis reducing the negative effects on wound healing potentially lowering the incidence of AL.

Design: This is a prospective, international, non-randomized, multicentre study.

Endpoints: The Primary objective of this trial is to assess the incidence of AL within 30 days after surgery. Secondary objectives are to assess anastomotic integrity at 90 days and 1 year, intraoperative efficacy and efficiency of the C-REX device, time to evacuation of the anastomotic ring, mode of evacuation and related patient experience, postoperative morbidity and readmissions, C-reactive protein (CRP) profile in the early postoperative period, functional outcomes, cost-effectiveness and surgical quality.

Population: A total of 165 patients (age ≥ 18 years) with histologically proven cT1-4aN0-2M0 cancer of the sigmoid colon or proximal rectum, or premalignant lesions not amenable to endoscopic resection, that require elective AR will be enrolled throughout 10 European colorectal centers.

Study procedures: The anastomosis will be created using the C-REX RectoAid Cath. The healing period will be approximately 10 days. The anastomotic ring detaches via necrosis and is evacuated with the feces. Patients will be asked to fill out questionnaires regarding Low Anterior Resection Syndrome (LARS) and use of healthcare and these will be gathered preoperatively, 90 days postoperative and 1 year after surgery. At 12 months a CT-scan and colonoscopy will be performed.

DETAILED DESCRIPTION:
Detailed description of device and surgical procedure:

During the surgical procedure, the colorectal anastomosis will be created using the C-REX RectoAid Cath (Carpo Novum AB, Halmstad, Sweden). The C-REX devices are CE-marked and used in its intended purpose in this trial. The C-REX RectoAid Cath is a refined anastomotic device that facilitates the construction of an inverted serosa-to-serosa adaptive colorectal anastomosis where the bowel ends are held together by snap-locking a proximal and distal silicone anastomotic ring. The C-REX devices can be used in both open and minimally invasive procedures. The proximal limit for C-REX RectoAid Cath is 25 cm above the anal verge and the distal limit is formed by the anal ring.

The anterior resection using the C-REX RectoAid Cath is performed by experienced colorectal surgeons who received training to use the C-REX device from an experienced Clinical Field Trainer from Carpo Novum AB. After bowel resection and measuring of the lumen using the C-REX Test Device, the proximal ring is placed using the C-REX LapAid. This device ensures that the colonic wall is folded around the anastomotic ring. Once this colonic ring is in position, the anvil is connected whereby catheters are placed into the colonic lumen. Subsequently, the C-REX RectoAid can be inserted transanal. In similarity to ordinary stapler devices, a concealed trocar becomes visible by rotating the knob on the base of the handle of the C-REX RectoAid. When possible, the stapler line of the transected proximal rectal stump is invaginated into the distal anastomotic C-REX ring and thus removed at firing of the RectoAid instrument. The trocar and proximal anvil are connected and by turning the knob clockwise, the gap between the anvil and the head of the instrument is closed. After firing the device, the two anastomotic rings are connected and the anastomosis is created. The four integrated catheters will be extracted simultaneous with the RectoAid instrument and can be used to measure the Anastomotic contact pressure (ACP) to validate the anastomosis. These catheters are in direct contact with the anastomotic healing site. When the anastomotic rings detach during the healing process by necrosis, after approximately 10 days, the anastomotic ring loosens from of the intestinal wall and is expelled with the feces.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven cancer of the sigmoid colon or proximal rectum (cT1-4aN0-2M0) that require AR as the procedure of choice or premalignant lesions not amenable to endoscopic resection, that require AR as the procedure of choice.
* Suitable for curative AR
* Suitable for elective laparoscopic or robotic surgery
* Cognitive ability to take part in the study, to understand the information the patient receives about participating in the study, to provide informed consent and to agree to complete the questionnaires.

Exclusion Criteria:

* Pre-existing health conditions requiring emergency surgery, such as intestinal obstruction or perforation, local or systemic infections, peritonitis, or intestinal ischemia.
* Cancer with distant metastases (TNM Stage IV).
* Intestinal or anal stenosis or other obstructions distal to the planned anastomosis.
* Prior pelvic radiation including neoadjuvant chemoradiotherapy.
* Contraindications to general anaesthesia.
* Need for defunctioning ileostomy (intention to treat).
* Patients who have a contra-indication for or are unable to receive preoperative bowel preparation or at least two enemas prior to surgery.
* Immunocompromised patients e.g. taking steroids or receiving immunotherapy.
* Any condition that, in the opinion of the investigator, may interfere with the study conduction. In particular, any condition which can cause significant alteration of colonic wall thickness such as chronic and repeated infection (e.g. diverticulitis) which may impair the use of C-REX RectoAid Cath

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 165 Patients (age ≥ 18 years) with histologically proven cT1-4aN0-2M0 cancer of the sigmoid colon or proximal rectum, or with premalignant lesions not amenable to endoscopic resection, that require AR as the procedure of choice
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage rate | 30 days
  The primary endpoint of clinical anastomotic leakage (AL) is defined, according to the International Study Group definition, as a confirmed defect of the intestinal wall at the ananstomotic site leading to a communication between the intra- and extraluminal compartments. Diagnosis of AL is made by either CT scan, flexible endoscopy or found at time of a reoperation. An abscess or collection of fluid in close proximity to the anastomosis will be deemed as an AL.

SECONDARY OUTCOMES:
Anastomotic leakage rate | 90 days
  Clinical anastomotic leakage is defined according to the International Study Group definition, as a confirmed defect of the intestinal wall at the ananstomotic site leading to a communication between the intra- and extraluminal compartments, within 90 days after surgery. Diagnosis of AL is made by either CT scan, flexible endoscopy or found at time of a reoperation. An abscess or collection of fluid in close proximity to the anastomosis will be deemed as an AL.
Anastomotic leakage rate | 1 year
  Clinical anastomotic leakage is defined according to the International Study Group definition, as a confirmed defect of the intestinal wall at the ananstomotic site leading to a communication between the intra- and extraluminal compartments, within 1 year after surgery. Diagnosis of AL is made by either CT scan, flexible endoscopy or found at time of a reoperation. An abscess or collection of fluid in close proximity to the anastomosis will be deemed as an AL.
Postoperative complications | 30 days
  Postoperative complications will be classified according to the Clavien-Dindo scale. The Clavien Dindo Classification is used to rank the severity of a surgical complication. It is based on the type of therapy needed to correct the complication. The scale consists of several grades (Grade I, II, IIIa, IIIb, IVa, IVb and V). A grade I complication is any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions whilst a Grade IV complication is a life-threatening complication requiring ICU-management.
Days until evacuation of the anastomotic ring | 14 days
  An anastomotic ring remains at the site of the anastomosis for approximately 10 days. The ring detaches via necrosis on the inner part of the intestinal surface and is evacuated with the feces. When the patient has not evacuated the ring after 14 days, the ring will be manually removed.
Number of readmissions | 90 days
  Any unplanned readmission within 90 days after surgery will be registered. Data will be derived from the electronic patient dossier.
Economical evaluation | 1 year
  An economical evaluation of the adaptive anastomosis technique will be performed. To ensure a broad evaluation of costst both direct costs will be collected using the iMTA Medical Consumption Questionnaire (iMCQ) as well as indirect costs such as production losses using the iMTA Productivity Cost Questionnaire (iPCQ). A combination of these two questionnaires combined with data from the patient file such as hospital stay and complications to determine direct medical costs will ensure a complete economical evaluation.
LARS score for functional outcomes | 1 year
  Measured by the internationally validated Low Anterior Resection Syndrome (LARS) score questionnaire. The questionnaire is composed of 5 questions that centre on the symptoms experienced by patients; the sum of all the items varies from 0 to 42 points, for classification into 3 groups: non-LARS (0-20 points), minor LARS (21-29 points) and major LARS (30-42 points). Patients will fill in the questionnaires before surgery, 90 days after surgery and 1 year after surgery
Surgeon satisfaction | Intraoperative
  Satisfaction with the performance and usability of the C-REX device is measured using the following questions:
  Overall satisfaction: (Very unsatisfied/unsatisfied/neutral/satisfied/very satisfied) Satisfaction with method of creation proximal anvil: (Very unsatisfied/unsatisfied/neutral/satisfied/very satisfied) Satisfaction with ring connection 'Stapling': (Very unsatisfied/unsatisfied/neutral/satisfied/very satisfied)
NASA Task Load Index | Intraoperative
  Though not mandatory, all surgeons are asked to fill out the NASA Task Load Index after surgery. Hart and Staveland's NASA Task Load Index method assesses work load on seven (Mental Demand, Physical Demand, Temporal Demand, Performance, Effort, Frustration) scales ranging from low (1) to high (20).
Serial CRP | 2-4 days
  Measured C-reactive protein (mg/l) in the early postoperative period (day 2-4).

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided